CLINICAL TRIAL: NCT06270732
Title: Efficacy of iMentalize and Mediational Intervention for Sensitizing Caregivers - Self Administered Version (MISC-SA) to Foster Parents' Mentalization and Children Mental Health in Families From General Population (iMentalize Project).
Brief Title: Efficacy of iMentalize and MISC-SA to Foster Parents' Mentalization and Children Mental Health in General Population.
Acronym: iMentalize
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Autonoma de Barcelona (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Principal Investigator, Sergi Ballespí, Ph.D., Principal Investigator, Universitat Autonoma de Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PID2021-125444OB-100-II-iM
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Emotional Intelligence; Social Interaction; Mental Health Wellness 1; Well-Being, Psychological
Keywords: Mentalization; Reflective function; Reflective parenting; Environmental enrichment; Parent-child interaction; Development; Mental Health; Emotional Health; Emotional well-being
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Double-blind, parallel group, randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental: iMentalize Program (iMentalize) (Experimental): iMentalize is a structured new program specifically designed to foster mentalization in non-clinical general population. Inspired in Mentalization Based Treatments, which foster mentalization as a principal factor for salutogenesis in clinical settings, iMentalize aims to promote the parents' mentalization stance by using 30 structured sessions where parents are trained in MISC components (Mediational Intervention for Sensitizing Caregivers) to specifically help children to mentalize about cartoon's characters, about themselves, about the caregiver's mental states and about other close others. iMentalize is administered to parent-child dyads who work together in weekly 45-minutes sessions across 1 year.
  Interventions: Behavioral: iMentalize Program (iMentalize)
- Mediational Intervention for Sensitizing Caregivers, Self-Administered (MISC-SA) (Experimental): This MISC version (MISC-SA) aims to transfer the MISC original training to wider communities by diminishing the cost of the teaching and learning. By implementing the MISC lessons in an online platform, thus allowing self-learning, the new Self- Administered version of MISC allows to obtain MISC training in 30 weekly sessions distributed across 12 months, in 2 blocks: 18 sessions from February to June, and 12 additional sessions from October to December. In contrast to the original version of MISC, this version allows the simultaneous self-training of a high number of participants with very low intervention of a supervisor, which diminishes the cost. MISC-SA keeps the core component of MISC training (video-feedback) by fostering participants to record interactions and then visualize them using guided reﬂection.
  Interventions: Behavioral: Mediational Intervention for Sensitizing Caregivers, Self-Administered version (MISC-SA)
- Mediational Intervention for Sensitizing Caregivers - Readings (MISC-R): Treatment as Usual (TAU) (Active Comparator): MISC-R is a more theoretical version of MISC training lacking the core MISC component (video-feedback). MISC-Readings provides the theoretical knowledge of MISC but lacking practice and reﬂection about MISC components by watching one's own video recorded interactions with the child. MISC-Readings substitutes all the time for practice and video-feedback with theoretical pills and readings, that is, with theoretical knowledge. Thus, this more theoretical MISC version can be assimilated to common intellectual trainings based on "cognitive" knowledge and pencil-and-paper exercises instead of skill-based training based on true practice for social-emotional skills development.
  Interventions: Behavioral: Mediational Intervention for Sensitizing Caregivers - Readings version (MISC-R): Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: iMentalize Program (iMentalize) — This is a 30-hour group training involving 30 sessions lasting 45 minutes and 7.5 hours of inter-sessions work.
  Session 1: Program presentation; Session 2: Reflective Parenting; Session 3: Cartoon's session I (baseline); Session 3: What is Mentalization; Session 4: Fundamentals of Human Interaction; Session 5: Cartoon's session II (the beginnings); Session 6: Mentalization and Mental Health; Session 7: MISC context and cultural components; Session 8: Cartoon's session III (practice with MISC context comp.); Session 9: The importance of emotions in human interaction; Session 10: MISC emotional components; Session 11: Cartoon's session IV (practice with emotional comp.); Session 11: How mentalization is developed; Session 12: MISC cognitive components; Session 13: Cartoon's session V (practice with cognitive comp.); Session 14: How to foster children mentalization skills. Sessions 15 to 30: Cartoon's sessions using MISC components to foster children mentalization.
  Other Names: iMentalize
  Arms: Experimental: iMentalize Program (iMentalize)
Behavioral: Mediational Intervention for Sensitizing Caregivers, Self-Administered version (MISC-SA) — This is a 30-hour individual training involving 30-weekly online, individual, self-administered 45' sessions (22.5h) + 7.5h of between sessions work (readings, supervision, video- recordings for later video-feedback, reﬂection exercises). BLOCK I: Session 1: Presentation of the MISC program; Sessions 2 to 8 (Self-Administered or SA): Theoretical bases of the MISC; Sessions 9-18 (MISC practice and video-feedback); Summer break: Recording daily life interactions; BLOCK II: Session 19: Recap; Sessions 20-30: guided reﬂection and video-feedback.
  Other Names: MISC-SA
  Arms: Mediational Intervention for Sensitizing Caregivers, Self-Administered (MISC-SA)
Behavioral: Mediational Intervention for Sensitizing Caregivers - Readings version (MISC-R): Treatment as Usual (TAU) — This is an equivalent 30-hour online self-administered training involving 30 x 45' individual online sessions (22.5h), mostly based on reﬂection exercises around brief readings, pills, and animated shorts, but not video- feedback and guided practice. This is complemented with 7.5h of between-sessions work based on looking for new information, adult-child (non-guided) activities (and not for later video- feedback) or out-of-line guided reﬂective exercises.
  Session 1: Program presentation; Session 2-8: Theoretical bases of MISC and mentalization; Session 9-16: MISC and mentalization applied to mental health; 17-18: Benefits of MISC to improve children learning; 19-20: Benefits of MISC for self-esteem; 21-22: The importance of MISC to foster mentalization; 23-24: Mentalization and pro-social behavior; 25-26: The importance of MISC to promote secure attachment; 27: MISC impact in epistemic trust; 28-29: MISC and well-being; 30: MISC, mentalization and environmental enrichment.
  Other Names: MISC-R, TAU
  Arms: Mediational Intervention for Sensitizing Caregivers - Readings (MISC-R): Treatment as Usual (TAU)

SUMMARY:
OBJECTIVES: The goal of this parallel randomized controlled trial is to test the efﬁcacy of the iMentalize program and the Mediational Intervention for Sensitizing Caregivers - Self Administered version (MISC-SA) to foster parents' mentalization and children mental health in families from general population.

PARTICIPANTS will randomly receive one of the 3 interventions, all based in 30 weekly online non-synchronic sessions extended across 1 year: the iMentalize program (based on parent-child sessions where they see and talk about cartoon shorts), the MISC-SA (self-administered MISC version based on guided video-feedback using recordings of one's own parent-child interactions), and MISC-R (also self-administered but mainly based on readings and cognitive exercises instead of video-feedback), which is used here as Treatment as Usual (TAU, control group) because it is the most similar to most other intellectual and mainly theoretical trainings.

COMPARISONS: Researchers will compare all 3 groups among them to see to what extent:

* iMentalize program shows efficacy in fostering mentalization compared with MISC-SA and TAU (control group).
* iMentalize program shows efficacy in fostering children's mental health compared with TAU (control group).
* MISC-SA shows efficacy in fostering parent's mentalization and children mental health compared with TAU (control group).

DETAILED DESCRIPTION:
CONTEXT: Mental health interventions are mostly provided once mental health is lost, that is, in context of psychopathology (i.e., when clinical levels of severity or impairment are reached). James Heckman's Equation suggests that investing in mental health before it is severely impaired would lead to high returns. We want to test: 1) to what extent is possible to transfer active ingredients for mental health from the clinical context to the community, and 2) to what extent an intervention aimed to enrich parents with higher mentalization and interaction skills improves children's mental health. Because this intervention aims to reach a wide community in non-clinical settings, it should be extensive (to ensure solid changes in the child environment) and cost-efﬁcient, that is: cheaper than those individually transmitted in the classic therapist-client relationship.

METHODOLOGY: 12-month multisite, Randomized, Controlled Trial (RCT).

MEASURES OPERATIONALIZATION: It is expected that this translational intervention which aims to move factors for salutogenesis from the clinical setting to the non-clinical range of the mental ill-health continuum could beneﬁt both the caregivers (parents) who receive the intervention and their children, who are daily exposed to them. Caregivers' beneﬁts are expected in terms of improved mentalizing capacities (primary outcome) but also in terms of higher quality interactions, lower stress, lower distress symptoms, higher well-being and higher sense of self- efﬁcacy (secondary outcomes). Child's mental health (primary outcome) is operationalized as multidimensional using: the number of symptoms, the level of role- and social functioning, and well-being. Child's beneﬁts in terms of mentalization and pro-social behavior (secondary outcomes) are also expected because of the long-term exposition to adults enriched with new social-emotional skills based on the intervention. It is expected that parent's interventions could foster children mental health by promoting children mentalization skills (mediational or process variable).

STATISTICAL ANALYSES: The analysis under the Intention-To-Treat (ITT) approach will encompass all participants subjected to random allocation, with the utilization of multiple imputation techniques to address any missing data. Estimation of parameters, accounting for the speciﬁc statistical assumptions of each model and the data's characteristics, will be carried out through the implementation of Linear Mixed-Effect Models and Structural Equation Modeling (SEM). Various R packages will be employed to execute these models, primarily "lme4" and "nlme" for linear mixed-effect models, and "lavaan" for SEM models. Concerning statistical power, a sample size of 105 participants (35 per arm) has been proposed, which exceeds the minimum of 54 participants (18 per arm) required to detect a medium effect size (Cohen's d=0.25) in the design comprising 3 arms, 3 repeated measures (pre, post, and 1 follow-up), and a power level of .95. An empirical power close to 1.00 is anticipated. Effect size measures, including Cohen's d and squared Omega statistics, will be employed.

ELIGIBILITY:
Inclusion Criteria:

* Parent of a 6 to 18 years old child
* Written informed consent
* Understanding Catalan
* Pre-intervention assessment complete

Exclusion Criteria:

* None

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2025-02-21 (Estimated); Study Completion 2025-03-03 (Estimated)

PRIMARY OUTCOMES:
Parental Reﬂective Function Questionnaire (PRFQ) | Through study completion, an average of 12 months
  This scale assesses parent capacity to mentalize the child (to keep the child's mind in mind) using 18 items scored from 1 (Completely disagree) to 7 (Completely agree). Total score ranges from18 to 126. A higher score indicates higher reﬂective parenting (better outcome).
Trait Meta-Mood Scale (24 items) (TMMS-24) | Through study completion, an average of 12 months
  This instrument consists of 3 x 8-tiem subscales ('attention to emotions', 'emotional clarity' and 'emotional repair') scored with a 5- point scale ranging from "1=totally disagree" to "5=totally agree". Each scale ranges 8-40. A higher score means higher meta- mood knowledge (better outcome).
Basic Empathy Scale (BES) | Through study completion, an average of 12 months
  This is a gold standard to assess empathy and consists of 20 items scored from 1 (totally disagree) to 5 (totally agree). Total score ranges from 20 to 100. A higher score is indicative of higher empathy (better outcome).
Movie for the Assessment of Social Cognition (MASC) | Through study completion, an average of 12 months
  The MASC consists of a 15-minute video stopping in 46 segments or items to assess adequate mentalizing, hyper-mentalizing, hypo-mentalizing or non-mentalizing. All scales range from 0 to 46. A higher score in adequate mentalizing indicates higher mentalizing capacity (better outcome). A higher score in the other 3 subscales indicates worse mentalizing capacity.
Stirling Children's Wellbeing Scale (SCWBS) | Through study completion, an average of 12 months
  This is a 15-item scale commonly used to measure children's happiness in the last 2 weeks. Items are scored from 1 (Never) to 5 (all the time). The score ranges from 15 to 75. A higher score means more happiness (better outcome).
Child Well-Being Level (CWBL) | Through study completion, an average of 12 months
  This is Lickert's 7-point scale to assess the child's level of happiness compared with other children of the same age. It ranges from '1=very less happy' to '8=very happier'. A higher score means more happiness (better outcome).
Strengths and Difﬁculties Questionnaire (SDQ) | Through study completion, an average of 12 months
  This is a 25 item-based scale, scored using a 3-points scale (0=not true; 2=certainly true) which provides a screening of 5 dimensions: children emotional problems, conduct problems, hyperactivity, peer-problems and pro-social behavior. All scales range from 0 to 10. A higher score means more problems (ﬁrst 4 scales: worse outcome) or more pro-social behavior (last subscale: better outcome).
Achenbach System for Empirically Assessment (ASEBA) | Through study completion, an average of 12 months
  This is a very well-known 110 items-based instrument scored from 0=Not true to 2=Very often true which provides a screening in 8 clinical dimensions and 3 second order scales. Each scale has a different range. Higher scores mean higher severity of mental health problems (worse outcome).

SECONDARY OUTCOMES:
Observing Mediational Interaction (OMI) | Through study completion, an average of 12 months
  This is the observational measure used in the Mediational Intervention for Sensitizing Caregivers (MISC) and quantiﬁes emotional (attachment-based) and cognitive (learning-based) behaviors during caregiver-child interaction. The emotional components scale ranges from 0 to 40. A higher score indicates more emotional components. Cognitive components (Focusing, Affecting, Expanding, Regulating, Rewarding) are evaluated based on their frequency along the interaction. A higher score means more frequency of those components (better outcome).
Parental Stress Questionnaire (PSI) | Through study completion, an average of 12 months
  This instrument consists of 36 items scored from 1 (very agree) to 5 (very disagree). Total score ranges from 36 to 180. A higher score indicates more parental stress (worse outcome).
Goldberg Health Questionnaire (28 items) (GHQ-28) | Through study completion, an average of 12 months
  This is a gold standard screening of adult psychopathology in 4 areas (anxiety, depression, somatic complaints, and social dysfunction). Each area is evaluated with 7 scores from 1 to 4. Subscales range from 7 to 28. A higher score indicates a higher level of problems (worse outcome).
Difﬁculties in Emotional Regulation Scale (DERS) | Through study completion, an average of 12 months
  This is a gold standard to assess problems of Emotional Regulation (a key factor for mental health) using 36 items with 5 response options ranging from "1=almost never" to "5=almost always". Total score ranges 36-180. A higher score means higher emotional regulation difﬁculty (worse outcome).
Oxford Happiness Questionnaire (OHQ) | Through study completion, an average of 12 months
  This is a gold standard to assess emotional well-being based on 8 items scored from "1=totally disagree" to "6=totally agree". The scale ranges from 8 to 48. A higher score indicates higher well-being (better outcome).
Rosenberg's Self-Esteem Scale (RSES) | Through study completion, an average of 12 months
  This is a gold standard to self-report adult self-esteem with 10 items scored from "1=totally agree" to "4=totally disagree". Total score ranges from 10 to 40. Once inverted, a higher score indicates higher self-esteem (better outcome).
Parental Sense of Competence Scale (PSOC) | Through study completion, an average of 12 months
  This scale consists of 10 items scored from 1 (totally disagree) to 6 (totally agree) to assess parental perceive self-competence. It ranges from 10 to 60. A higher score indicates a higher sense of self-competence in parenting (better outcome).
Self-Other Mentalization Scale (SOMS) | Through study completion, an average of 12 months
  This is a 10 items-based scale answered from 1 (very less than others) to 5 (much more than others). Self- and Other- subscales scores range from 5 to 25. Higher scores mean higher mentalization capacity (better outcome)
Reﬂective Functioning Scale - Youth (5 items version) (RFQ-Y5) | Through study completion, an average of 12 months
  This is a shorter version of Fonagy's Reﬂective Function Questionnaire. It includes 5 items scored from 1 (very disagree) to 5 (very agree) and ranges from 5 to 25, being a higher score indicative of higher mentalization capacity (better outcome).
Trait Meta-Mood Scale - Children version (TMMS-C) | Through study completion, an average of 12 months
  This instrument is here used as a measure of self-mentalizing. Only the 5 item-scale of 'clarity of emotions' will be used. Items score from 1=Not at all true, to 5=Completely true. Total score ranges from 5 to 25, being a higher score indicative of higher emotional clarity (better outcome).
Big Five Questionnaire for Children and Adolescents (BFQ-NA) | Through study completion, an average of 12 months
  This questionnaire assesses the big ﬁve personality factors in young children using 65 items scored from 1=Almost always to 5=Almost never. In this study, the scale of kindness is used to score pro-social behavior, and the scale of emotional instability to score emotional dysregulation. A higher score indicates higher emotional instability (worse outcome) or higher pro-sociality (better outcome, after inverting the score).
BarOn Inventory of Emotional Intelligence for children aged 7 to 18 years old (BarOn) | Through study completion, an average of 12 months
  BarOn's scales of intra-personal (6 items) and inter-personal (12 items) scales, which are scored in 4-points scales ranging from '1=Never' to '4=Always'. The indicated subscales ranges are 4-24 and 12-48, respectively. A higher score indicates higher intelligence (better outcome).
Rosenberg's Self-Esteem Scale - Child version (RSES-C) | Through study completion, an average of 12 months
  This is a gold standard measure of self-esteem using 10 items which scored from "1=totally agree" to "4=totally disagree". After inverting the total score, which ranges from 10 to 40, a higher score means higher self-esteem (better outcome).
Battery of Socialization (BAS) | Through study completion, an average of 12 months
  The scales of social sensitivity, respect and self-control, and aggressivity, all scored using items ranging from Never (1) to Always (4), are here used to measure children's pro-social behavior. Higher scores mean higher pro-social dimensions (better outcome).

OTHER OUTCOMES:
Inventory of Learning Patterns, reduced version (60 items) (ILP-60) | Through study completion, an average of 12 months
  This instrument measures learning patterns, which are considered to moderate the impact of the intervention. It consists of 60 items evaluating 4 learning components (processing strategies, regulation strategies, conceptions of learning, learning orientations) with 15 x 5-point Lickert scale items each. All scales range from 15 to 75. A higher score means a higher presence of that component or a higher tendency to use that pattern (potential moderator).
Relationship Questionnaire (RQ) | Through study completion, an average of 12 months
  This is a very brief screening scale including 4 x 7-point Lickert's to assess the 4 Bartholomew and Horowitz's relationship styles (secure, anxious-avoidant, anxious-preoccupied and disorganized) and 1 last categorical item to select the style that better identiﬁes the participant. Attachment style could moderate the impact of parental intervention on a child's mental health. Each attachment style is scored from 1 to 7. A higher score indicates a higher presence of that relationship style (potential moderator).
Time with the Child (TC) | Through study completion, an average of 12 months
  This is an ad hoc scale to calculate the amount of real time of interaction (communication and reciprocal influence) with the child in daily minutes, across 1 week (from Monday to Sunday). It ranges from 0 to several hours. A higher score means more time for real interaction with the child (in minutes) per day or per week. This is used as a measure of exposure to the "enriched" parenting (potential moderator).

CONTACTS AND LOCATIONS:
Overall Officials: Sergi Ballespí, Researcher, Principal Investigator — Universitat Autònoma de Barcelona
Locations (2):
- Spain (2):
  - Sergi Ballespí, Barcelona
  - Universitat Autònoma de Barcelona, Barcelona

IPD SHARING:
Plan to Share IPD: No
The base of data will be shared through Universitat Autònoma de Barcelona (UAB) public repository.

REFERENCES:
- See also: Mentalization and Mental Health Laboratory — http://www.mamhlab.cat/
- See also: Heckman Curve — https://heckmanequation.org/resource/the-heckman-curve/